CLINICAL TRIAL: NCT01988350
Title: Pancreatic Insufficiency Secondary to Tobacco Exposure
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Field Willingham MD, Director of Endoscopy, Emory University
Other Study IDs: IRB00064360
Record Dates: First submitted 2013-07-24; First posted 2013-11-20 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Pancreatic Insufficiency
Keywords: pancreatic insufficiency; pancreatic elastase; fecal elastase; smoking; tobacco
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-smokers
- Smokers

SUMMARY:
Pancreatic insufficiency is a condition in which there is a decrease in the production and release of enzymes made in the pancreas, which causes nutrient malabsorption. There are many chronic diseases that can lead to pancreatic insufficiency. In the early stages of this disease, a patient may not experience any symptoms, and the prevalence of pancreatic insufficiency may be underestimated. Smoking has long been recognized as a cause of disease in many organs in the body. Cigarette smoke causes inflammation and damages tissue, including the pancreas. Studies have shown that smoking is an independent risk factor for pancreatic cancer and chronic pancreatitis. It has also been shown that the more a person smokes, the worse his disease will be. Additionally, there are studies that show that smokers have nutritional deficiencies. There are observational and retrospective studies that suggest that pancreatic insufficiency may also be caused by smoking. However, this has not been established, and the relationship has not been examined in a controlled manner. This study examines the relationship between smoking and pancreatic insufficiency in patients who do not have other pancreatic diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 30 years of age
2. Able to read, understand, and sign informed consent
3. Patients with a negligible smoking history (defined as no smoking for the past 7 years, and a total smoking history ≤ 5 pack-years) OR patients with AT LEAST a 20 pack-year smoking history

Exclusion Criteria:

1. Patients with a prior diagnosis of pancreatic insufficiency
2. Patients who have a current or remote history of acute or chronic pancreatitis or any other primary pancreatic disease or malignancy
3. Patients who have had pancreatic surgery
4. Patients with a diagnosis of small bowel malabsorption or Celiac disease
5. Patients with any other significant systemic disease that is deemed by the investigator as possibly interfering with the conduct or interpretation of the study

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Smokers and non-smoking controls without a h/o pancreatic disease.
Sampling Method: Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
pancreatic insufficency | 1-2 weeks after provision of stool specimen
  The primary outcome is presence or absence of pancreatic insufficiency as determined by fecal elastase-1 measurement

CONTACTS AND LOCATIONS:
Overall Officials: Field F Willingham, MD, MPH, Principal Investigator — Emory University School of Medicine, Division of Gastroenterology
Locations (1):
- The Emory Clinic, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Raphael KL, Chawla S, Kim S, Keith CG, Propp DR, Chen ZN, Woods KE, Keilin SA, Cai Q, Willingham FF. Pancreatic Insufficiency Secondary to Tobacco Exposure: A Controlled Cross-Sectional Evaluation. Pancreas. 2017 Feb;46(2):237-243. doi: 10.1097/MPA.0000000000000721. PMID 27846134